CLINICAL TRIAL: NCT01056809
Title: Treatment Strategies for Primarily Generalized Colorectal Cancer Prospective Randomized Comparison Between Two Treatment Strategies
Brief Title: Treatment Strategies for Primarily Generalized Colorectal Cancer
Acronym: PGC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too slow recruitment
Sponsor: Vrinnevi Hospital (Other)
Collaborators: Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Principal Investigator, Gunnar Arbman, Consultant surgeon, Vrinnevi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGC-8
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Metastases; Treatment strategies; Colorectal cancer with synchronous metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional strategy (Active Comparator): First resection of the primary colorectal tumour, then treatment of metastases with chemotherapy and if possible surgery.
  Interventions: Procedure: Chemotherapy and surgery
- Alternative strategy (Active Comparator): First treatment of metastases with chemotherapy and if possible surgery, later resection of primary colorectal tumour if hope for cure or if symptoms develope that necessitates treatment
  Interventions: Procedure: Chemotherapy and surgery

INTERVENTIONS:
Procedure: Chemotherapy and surgery — Treatment not specified but in accordance with national guidelines

SUMMARY:
For patients with primarily generalized colorectal cancer two treatment strategies are compared to establish which strategy gives best overall survival.

The traditional strategy is to first resect the primary colorectal tumour and then treat the metastases with chemotherapy followed if possible by surgery.

The alternative strategy is to first treat the metastases with chemotherapy followed if possible by surgery and only resect the primary colorectal tumour if there is hope for cure or if symptoms develop that necessitates treatment.

DETAILED DESCRIPTION:
Patients are randomized between the two treatment strategies mentioned above. After initial treatment the patients are categorized as palliative or treated with curative intent. Patients are followed with quality of life evaluations every 6 months. Outpatient visits, hospital care, examinations and treatment are recorded as well as complications and side effects. Survival is recorded and for those patients treated with curative intent the tumour situation 3 years after randomization is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primarily generalized colorectal cancer diagnosed by pathology or typical appearance on x-ray or at endoscopy and where there is uncertainty regarding best treatment strategy

Exclusion Criteria:

* Patients not willing to participate or unable to sign informed consent.
* Patients with other malignancy with metastatic potential
* Patients where synchronous resection of primary tumour and metastases is planned
* Patients not fit for chemotherapy or surgery
* Patients with locally unresectable primary tumours
* Patients with symptoms from primary colorectal tumour necessitating resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years after completion of study

SECONDARY OUTCOMES:
3 year survival for patients treated with curative intent | 3 years after randomization
Palliative patients not receiving chemotherapy treated with the traditional strategy | Completion of study
Quality of life | Every 6 months up to 3 years
Health care consumption | Completion of study
Complications and side effects | Completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Arbman, MD, PhD, Principal Investigator — Department of Surgery in Östergötland; Per Sandström, MD, PhD, Study Chair — Department of Surgery in Östergötland; Hans Starkhammar, MD, PhD, Study Chair — Regional Oncologic Center, Linköping; Bengt Glimelius, Professor, Study Chair — University of Uppsala, The Karolinska University Hospital, Stockholm; Lars Lundell, Professor, Study Chair — The Karolinska University Hospital, Stockholm; Per-Olof Nyström, Professor, Study Chair — The Karolinska Universtiy Hospital, Stockholm; Ulf Gunnarsson, Professor, Study Chair — The Karolinska University hospital, Stockholm; Lars Påhlman, Professor, Study Chair — Uppsala University
Locations (10):
- Sweden (10):
  - Höglandssjukhuset, Eksjö
  - Department of Surgery, Gävle - Hudiksvall
  - Länssjukhuset Ryhov, Jönköping
  - Länssjukhuset, Kalmar
  - Universitetssjukhuset, Linköping
  - Vrinnevisjukhuset, Norrköping
  - Karolinska Universitetssjukhuset, Stockholm
  - Akademiska sjukhuset, Uppsala
  - Värnamo sjukhus, Värnamo
  - Centrallasarettet, Västerås

REFERENCES:
- [Background] Mentha G, Majno PE, Andres A, Rubbia-Brandt L, Morel P, Roth AD. Neoadjuvant chemotherapy and resection of advanced synchronous liver metastases before treatment of the colorectal primary. Br J Surg. 2006 Jul;93(7):872-8. doi: 10.1002/bjs.5346. PMID 16671066
- [Background] Scoggins CR, Meszoely IM, Blanke CD, Beauchamp RD, Leach SD. Nonoperative management of primary colorectal cancer in patients with stage IV disease. Ann Surg Oncol. 1999 Oct-Nov;6(7):651-7. doi: 10.1007/s10434-999-0651-x. PMID 10560850
- [Background] Benoist S, Pautrat K, Mitry E, Rougier P, Penna C, Nordlinger B. Treatment strategy for patients with colorectal cancer and synchronous irresectable liver metastases. Br J Surg. 2005 Sep;92(9):1155-60. doi: 10.1002/bjs.5060. PMID 16035135
- [Background] Scheer MG, Sloots CE, van der Wilt GJ, Ruers TJ. Management of patients with asymptomatic colorectal cancer and synchronous irresectable metastases. Ann Oncol. 2008 Nov;19(11):1829-35. doi: 10.1093/annonc/mdn398. Epub 2008 Jul 28. PMID 18662955